CLINICAL TRIAL: NCT00589875
Title: A Phase IIa Study of AdV-tk + Valacyclovir Gene Therapy in Combination With Standard Radiation Therapy for Malignant Gliomas
Brief Title: Phase 2a Study of CAN-2409 With Standard Radiation Therapy for Malignant Glioma
Acronym: BrTK02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrTK02
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; Anaplastic Astrocytoma; High Grade Glioma
Keywords: Immunotherapy; Cytotoxicity; Tumor vaccine; CAN-2409; AdV-tk; Candel Therapeutics, Inc.
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma | interventions — Valacyclovir; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): This study is an extension of evaluation of the surgical resection arm, Arm B, from a phase Ib study in which dose escalation on arm B was completed.
  Interventions: Biological: CAN-2409; Drug: Valacyclovir; Drug: Temozolomide; Radiation: Radiation therapy

INTERVENTIONS:
Biological: CAN-2409 — Single dose of 3x10e11 vector particles of CAN-2409 delivered to the tumor bed after resection on day 0.
Drug: Valacyclovir — Single course of valacyclovir at dose of 2 grams orally three times per day for 14 days starting on day 1-3
  Other Names: Valtrex
Drug: Temozolomide — Concomitant TMZ will be administered orally once a day at a dose of 75 mg/m2 starting the next day after completing prodrug and continued for 6 weeks. Adjuvant TMZ will be administered days 1 to 5 of a 28-day cycle for 6 cycles with 150 mg/m2 administered for cycle 1, and 150 to 200 mg/m2 administered for cycles 2 to 6. Adjuvant treatment will start 1 month following completing RT.
Radiation: Radiation therapy — Radiation will be administered to up-front patients as per standard of care for the patient. It will start 3-7 days after CAN-2409 injection, preferably closer to 3 days. It will consist of standard external field radiation, limited to the area of tumor and brain adjacent to tumor, fractionated at doses of 200cGy per day for approximately 6 weeks to a total of 5500-6000 cGy.

SUMMARY:
The purpose of this study was to evaluate the safety and potential efficacy of CAN-2409 (also known / previously described as AdV-tk, GMCI) for malignant gliomas. The approach used an adenoviral vector (disabled virus) engineered to express the Herpes thymidine kinase gene (aglatimagene besadenovec, CAN-2409), followed by an antiherpetic prodrug, valacyclovir. CAN-2409 was injected into the resection bed after standard tumor surgery and valacyclovir pills were taken for 14 days. Standard radiation and chemotherapy were administered which have been shown to work cooperatively with CAN-2409 + prodrug to kill tumor cells. The hypothesis is that this combination therapy can be safely delivered and will lead to improvement in the clinical outcome for patients with newly diagnosed malignant gliomas, including glioblastoma multiforme (WHO grade IV) and anaplastic astrocytomas (WHO grade III).

DETAILED DESCRIPTION:
Patients had resectable or partially resectable malignant glioma and received injection of CAN-2409 into remaining tumor or tumor bed after resection. Pathologic confirmation of malignant glioma must be made prior to CAN-2409 injection; if this was not possible, the injection was not performed and the subject was no longer eligible for the study. The oral prodrug, valacyclovir, started 1-3 days after CAN-2409 injection and continued for 14 days. Standard radiotherapy began on average 7 days after CAN-2409 injection for the up-front course. Patients received temozolomide as per standard of care after completion of prodrug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have presumed resectable or partially resectable malignant glioma based on clinical and radiologic evaluation (pathologic confirmation of malignant glioma must be made at the time of surgery if not previously determined). Patients who have previously received CAN-2409 + prodrug on this study may receive an additional CAN-2409 + prodrug course at recurrence if eligibility criteria are still met.
* Tumor must be accessible for injection and must not be located in the brainstem, midbrain, contained within the ventricular system, or located in an infratentorial location.
* Upfront patients must be planning to undergo standard radiation therapy.
* Patients must be 18 years of age or older.
* Performance status must be KPS ≥70.
* Patients must have SGOT (AST) < 3x upper limit of normal.
* Patients must have serum creatinine < 2mg/dl and calculated creatinine clearance >10ml/min.
* Patients must have platelets > 100,000/mm3 and WBC > 3000/mm3.
* Patients of reproductive age must agree to use a medically accepted form of birth control while on the study.
* Patients must give study specific informed consent prior to enrollment. For re-administration, patients must be re-consented.
* Patients must be able to tolerate MRI scan procedure

Exclusion Criteria:

* Active liver disease including cirrhosis or hepatitis
* Patients on immunosuppressive drugs (with exception of corticosteroid)
* Known HIV+ patients.
* Patients with acute infections (viral, bacterial or fungal infections requiring therapy).
* Pregnant or breast feeding patients. Female patients of childbearing age must have negative serum or urine pregnancy test within 1 week of beginning therapy.
* Evidence of metastatic disease or other malignancy (except squamous or basal cell skin cancers).
* Other serious co-morbid illness or compromised organ function.
* Patients may not receive chemotherapy until valacyclovir is completed and may not receive other investigational anti-tumor agents within 30 days prior to study entry or during active participation in the study (defined as from CAN-2409 injection until tumor progression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-03; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Antonio Chiocca, MD, PhD, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - The University of Chicago, Chicago, Illinois
  - The Ohio State University Medical Center, Dept. Neurological Surgery, Columbus, Ohio
  - The Methodist Hospital Neurological Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wheeler LA, Manzanera AG, Bell SD, Cavaliere R, McGregor JM, Grecula JC, Newton HB, Lo SS, Badie B, Portnow J, Teh BS, Trask TW, Baskin DS, New PZ, Aguilar LK, Aguilar-Cordova E, Chiocca EA. Phase II multicenter study of gene-mediated cytotoxic immunotherapy as adjuvant to surgical resection for newly diagnosed malignant glioma. Neuro Oncol. 2016 Aug;18(8):1137-45. doi: 10.1093/neuonc/now002. Epub 2016 Feb 2. PMID 26843484
- See also: Phase II multicenter study of gene-mediated cytotoxic immunotherapy as adjuvant to surgical resection for newly diagnosed malignant glioma — https://pubmed.ncbi.nlm.nih.gov/26843484/

RESULTS

PARTICIPANT FLOW:
Period: Enrollment to Treatment Initiation
Arm/Group | Single Arm
Started | 52
Completed | 43
Not Completed | 9
Not completed — Patients ineligable for study. | 9
Period: Treatment Initiation to Completion
Arm/Group | Single Arm
Started | 43
Completed | 36
Not Completed | 7
Not completed — Treatment discontinuation | 7

BASELINE CHARACTERISTICS:
Population: All patient who initated experimental treatment in the study
Arm/Group | Single Arm
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants] — Population: 9 patients were withdrawn from the study prior to receiving treatment due to pathology inconsistent with malignant glioma.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 33
    >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 9 patients were withdrawn from the study prior to receiving treatment due to pathology inconsistent with malignant glioma.
  Participants
    Female | 13
    Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 9 patients were withdrawn from the study prior to receiving treatment due to pathology inconsistent with malignant glioma.
  Participants
    Hispanic or Latino | 6
    Not Hispanic or Latino | 37
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 9 patients were withdrawn from the study prior to receiving treatment due to pathology inconsistent with malignant glioma.
  Participants
    American Indian or Alaska Native | 0
    Asian | 2
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 41
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 43
Participants | 21

2. Secondary Outcome: Overall Survival
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm
Number analyzed (Participants) | 36
Months | 18.15 [13.60 to 25.00]

3. Other Pre Specified Outcome: Progression Free Survival
Time Frame: 24 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy - Brain (FACT-Br)
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to 2 months. All-Cause Mortality was assessed up to 5 years
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 41/43
Serious Adverse Events (participants affected / at risk) | 20/43
Other Adverse Events (participants affected / at risk) | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=43)
Arrhythmia (Cardiac disorders) | 1
Fever (General disorders) | 4
Dehydration (Gastrointestinal disorders) | 1
Pancreatitis (Hepatobiliary disorders) | 1
Wound Infection (Infections and infestations) | 1
Cerebral Edema (Nervous system disorders) | 3
Cognitive Disturbance (Nervous system disorders) | 2
Generalized Weakness (Nervous system disorders) | 1
Mood Alteration - Agitation (Nervous system disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 3
Fall (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Cystic Fluid Collection (Surgical and medical procedures) | 1
Thrombosis Embolism (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=43)
Tinnitus (Ear and labyrinth disorders) | 3
Fatigue (General disorders) | 22
Fever (General disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Anorexia (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 6
Taste Alteration (Gastrointestinal disorders) | 3
Urinary Tract Infection (Renal and urinary disorders) | 4
Edema (Blood and lymphatic system disorders) | 3
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5
Ataxia (Nervous system disorders) | 3
Cerebral Edema (Nervous system disorders) | 3
Cognitive Disturbance (Nervous system disorders) | 4
Memory Impairment (Nervous system disorders) | 7
Mood Alteration - Agitation (Nervous system disorders) | 3
Mood Alteration - Anxiety (Nervous system disorders) | 4
Mood Alteration - Depression (Nervous system disorders) | 9
Neuropathy - Motor (Nervous system disorders) | 5
Seizure (Nervous system disorders) | 11
Speech Impairment (Nervous system disorders) | 9
Headache (Nervous system disorders) | 21
Incision Site Pain (Surgical and medical procedures) | 3
Thrombosis Embolism (Vascular disorders) | 5
Insomnia (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No